CLINICAL TRIAL: NCT03355768
Title: Randomized Study of Romidepsin Versus the Combination of Romidepsin Plus Pralatrexate in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: Romidepsin Versus Combination of Romidepsin Plus Pralatrexate in PTCL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never opened due to lack of funding
Sponsor: Jennifer Amengual (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Amengual, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAR5550
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Romidepsin; Pralatrexate; PTCL; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — romidepsin; 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romidepsin Arm (Experimental): Control Arm: Subjects will receive Romidepsin 14 mg/m2 on Days 1, 8, 15.
  Interventions: Drug: Romidepsin
- Romidepsin + Pralatrexate Combination Arm (Experimental): Combination Arm: Subjects will receive Romidepsin 12 mg/m2 and Pralatrexate 25 mg/m2.
  Interventions: Drug: Romidepsin; Drug: Pralatrexate

INTERVENTIONS:
Drug: Romidepsin — Intravenous administration on a 28 day cycle
  Other Names: Istodax
Drug: Pralatrexate — Intravenous administration on a 28 day cycle
  Other Names: Folotyn
  Arms: Romidepsin + Pralatrexate Combination Arm

SUMMARY:
This study employs a 1:1 randomization of patients to receive romidepsin alone verses romidepsin plus pralatrexate for the treatment of patients with relapsed or refractory peripheral T-cell lymphoma (PTCL). The primary objectives will be to identify a 75% improvement in progression free survival (PFS) among patients receiving the combination compared to single agent romidepsin.

DETAILED DESCRIPTION:
Over the past 8 years, 3 new classes of drugs have been approved for the group of diseases recognized as peripheral T-cell lymphoma (PTCL). The novel anti-folate pralatrexate was the first drug approved for patients with relapsed or refractory PTCL in 2009. Four histone deacetylase (HDAC) inhibitors have been approved including vorinostat, romidepsin, belinostat, and chidamide (approved in China). The antibody drug conjugate Brentuximab vedotin was approved in one subtype of PTCL, anaplastic large T-cell lymphoma. The HDAC inhibitors and pralatrexate exhibit near lineage-specific activity with limited-to-no activity in B-cell lymphomas. As single agents in the relapsed setting romidepsin and pralatrexate exhibit response rates of 25-38% and 29-54% respectively across published phase I and II studies. While these studies are not identical in their patient composition, they included patients who are heavily pre-treated from a diversity of PTCL subtypes. A recent case match control analysis has demonstrated that patients treated with pralatrexate on PROPEL achieve a statistically significant survival advantage when compared to a matched historical population. In addition, sub-analysis of patients treated on PROPEL revealed that response and clinical benefit metrics (ORR, CR, duration of response (DOR) and progression free survival (PFS)) with pralatrexate improved significantly as the therapy moved up earlier in their treatment course. Patients achieving a response to romidepsin also exhibited a prolonged DOR of 28 months, with the median DOR not being reached in patients achieving complete response (CR).

The curative treatment of PTCL is not likely to be accomplished by the use of any single agent therapies. Clinically it makes sense to identify rational combinations of active agents in an attempt to identify disease specific active combinations. In preclinical models of T-cell lymphoma, in vitro cytotoxicity assays have clearly established a synergistic interaction between pralatrexate and several HDACI, including romidepsin. In addition, pralatrexate and romidepsin have differing mechanisms of actions and different toxicity profiles which lends to the probability that the combination of these agents will be combined safely with likely improved efficacy. Despite this rationale, the identification of a biological rationale will provide important insights into the optimal strategies for combing these different classes of drugs. It will also provide opportunities to develop biomarkers of response.

Peripheral T-cell lymphoma (PTCL) is extremely rare especially in the United States and Europe and is associated with considerable heterogeneity. Of the lymphomas, T-cell lymphomas make up a larger fraction in Asia and Latin America likely owing to genetic predisposition and early exposure to viral infections such as human T-lymphotropic virus type -1 (HTLV-1) and Epstein barr virus (EBV). Although there are differences between subtypes, in general patients with T-cell lymphomas have an inferior overall survival as compared to those with their B-cell lymphoma counterparts. The median overall survival of patients with T-cell lymphoma is only 1 to 3 years. There is presently no consensus on the best front-line therapy for these patients, though most recognize cyclophosphamide- doxorubicin hydrochloride (Adriamycin)-vincristine (Oncovin)-prednisolone (CHOP) or CHOP-based treatment as the standard despite the poor results. While clinical trials have been important in identifying novel agents active in relapsed disease, accrual to trials is often difficult given the rarity of the disease. Incorporation of novel agents into the front-line setting has not yet been realized.

Modest attempts to improve responses and duration of response have been made by intensifying front-line chemotherapy with the addition of etoposide and by consolidating response with autologous stem cell transplantation in the first remission, though these maneuvers have likely not significantly impacted the natural history of the disease.

Over the past several years, the investigators have adopted a strategy of trying to develop novel T-cell lymphoma active combinations, based on drug: drug synergy experiments in the preclinical setting. For example, the investigators have established biological preclinical and clinical evidence for the following doublets: (1) pralatrexate plus romidepsin (2) hypomethylating agents and HDAC inhibitors (3) pralatrexate plus gemcitabine.(4) pralatrexate plus bortezomib and (5) alisertib plus romidepsin. Each of these combinations leveraged a strong rationale for the companion agent used in combination with the HDAC inhibitor and or pralatrexate, leading to a clinical study in most cases.

Results from the phase I portion of the study demonstrate that the combination is safe and produces clinically meaningful responses across a diversity of PTCL subtypes in patients who are heavily treated. Twenty-nine patients were enrolled and were evaluable for toxicity. There were 3 dose-limiting toxicities (DLTs) in cohort 4 (pralatrexate 20mg/m2 & romidepsin 12mg/m2given weekly x 2 Q21D) consisting of 2 Grade 3 oral mucositis and 1 Grade 4 sepsis. The every other week (QOW Q28D) schedule had no DLTs at equivalent and higher doses. The grade 3/4 toxicities reported in >5% of patients included: neutropenia (28%), thrombocytopenia (28%), anemia (29%), oral mucositis (14%), hyponatremia (7%), pneumonia (7%) and sepsis (7%). Twenty-three patients were evaluable for response. The overall response rate (ORR) in the total, non-PTCL and PTCL populations was 57%; 33% (no CR) and 71% (40% CR) respectively. Given these are two approved agents for relapsed PTCL, there is a clear regulatory strategy following the completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed or refractory aggressive peripheral T-cell lymphoma as defined by 2016 World Health Organization (WHO) criteria (excluding nasal natural killer t-cell (NK-T) and blastic natural killer (NK))
* Patients are required to have no more than 5 lines of prior therapy (with cytoreductive therapy followed by autologous stem cell transplant counting as one line of therapy. Patients are eligible if they have relapsed after prior autologous or allogeneic stem cell transplant
* Measurable Disease
* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patients must have adequate organ and marrow function
* Adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior Therapy
* Prior exposure to pralatrexate or a histone deacetylase inhibitor (romidepsin, chidamide, belinostat, or vonrinostat)
* Exposure to chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs.
* No other concurrent investigational agents are allowed.
* Central nervous system metastases, including lymphomatous meningitis
* Uncontrolled intercurrent illness
* Pregnant women
* Nursing women
* Current malignancy or history of a prior malignancy
* Patient known to be Human Immunodeficiency Virus (HIV)-positive
* Active Hepatitis A, Hepatitis B, or Hepatitis C infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | up to 3 years
  Compare the progression free survival (PFS) in patients with R/R PTCL treated with romidepsin versus the combination of romidepsin plus pralatrexate.

SECONDARY OUTCOMES:
Complete Response (CR) | up to 3 years
  Contrast the complete response rate (CR) for patients treated with romidepsin or romidepsin plus pralatrexate.
Duration of response (DOR) | up to 3 years
  Contrast the duration of response (DOR) for patients treated with romidepsin or romidepsin plus pralatrexate.
Overall survival (OS) | up to 3 years
  Contrast the overall survival (OS)for patients treated with romidepsin or romidepsin plus pralatrexate.
Overall response rate (ORR) | up to 3 years
  Contrast the overall response rate (ORR) for patients treated with romidepsin or romidepsin plus pralatrexate.
Time to Treatment Progression (TTP) | up to 3 years
  TTP measured for patients with relapsed or refractory PTCL treated with romidepsin or romidepsin plus pralatrexate.
Time to Relapse (TTR) | up to 3 years
  TTR measured for patients with relapsed or refractory PTCL treated with romidepsin or romidepsin plus pralatrexate.
Maximum Number of Treatment Cycles | Up to 6 months
  Describe the maximum number of cycles and planned dose intensity of all drugs in both arms in patients with R/R PTCL treated with romidepsin or romidepsin plus pralatrexate.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Amengual, MD, Principal Investigator — Center for Lymphoid Malignancies Columbia University Medical Center